CLINICAL TRIAL: NCT00227838
Title: Modifying Group Therapy for Bipolar Abusers
Brief Title: Modifying Group Therapy for Bipolar Substance Abusers - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15968-1; R01-15968-1
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-09

CONDITIONS: Bipolar Disorder; Substance Dependence
Keywords: substance abuse
MeSH Terms: conditions — Bipolar Disorder; Substance-Related Disorders | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to modify Integrated Group Therapy (IGT), which is has been found successful for patients with bipolar disorder (BD) and substance use disorder(SUD), so that it can be more readily adopted by community drug abuse treatment programs. IGT is being reduced from 20 to 12 sessions in this trial, and is being conducted by front-line drug counselors, to test its effectiveness in a more community-based setting. The training has been expanded so that counselors without much psychopathology training or cognitive behavioral therapy experience can conduct IGT.

DETAILED DESCRIPTION:
IGT is being compared with 12 sessions of Group Drug Counseling (GDC) in a randomized controlled trial, with a sample size of 60 subjects. GDC is the type of treatment one would likely receive in a community drug abuse treatment program, in that it focuses primarily in substance use, unlike IGT, which focuses equally on SUD and BD issues. Patients are followed for a year after the end of the group therapy, to examine the long-term effects of the treatment, and also to examine the longer-term relationship of substance use and mood. Patients in the trial must be taking a mood stabilizer to enter the study. Any drug of abuse is accepted, and all subtypes of BD are accepted.

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder substance dependence taking a mood stabilizer

Exclusion Criteria:

* acute psychosis no substance use in past 60 days no prescribing doctor will not be in area for next 15 months lives too far away

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-07; Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Addiction severity

CONTACTS AND LOCATIONS:
Overall Officials: Roger Weiss, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Dept. of Psychiatry, Belmont, Massachusetts, United States

REFERENCES:
- [Derived] McDonald LJ, Griffin ML, Kolodziej ME, Fitzmaurice GM, Weiss RD. The impact of drug use in social networks of patients with substance use and bipolar disorders. Am J Addict. 2011 Mar-Apr;20(2):100-5. doi: 10.1111/j.1521-0391.2010.00117.x. Epub 2011 Feb 1. PMID 21314751
- [Derived] Weiss RD, Griffin ML, Jaffee WB, Bender RE, Graff FS, Gallop RJ, Fitzmaurice GM. A "community-friendly" version of integrated group therapy for patients with bipolar disorder and substance dependence: a randomized controlled trial. Drug Alcohol Depend. 2009 Oct 1;104(3):212-9. doi: 10.1016/j.drugalcdep.2009.04.018. Epub 2009 Jul 1. PMID 19573999
- [Derived] Jaffee WB, Griffin ML, Gallop R, Meade CS, Graff F, Bender RE, Weiss RD. Depression precipitated by alcohol use in patients with co-occurring bipolar and substance use disorders. J Clin Psychiatry. 2009 Feb;70(2):171-6. doi: 10.4088/jcp.08m04011. Epub 2008 Dec 30. PMID 19192456